CLINICAL TRIAL: NCT04074499
Title: What Daily Activities Increase the Risk of Falling in Chronic Obstructive Pulmonary Disease Patients?
Brief Title: The Risk of Falling in Patients with Chronic Obstructive Pulmonary Disease
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, MSc Research Assistant, Istanbul University - Cerrahpasa
Other Study IDs: 459535
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Fall; Balance; Distorted; Activity, Motor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group-1: The patients were classified based on the frequency of falls in the last 12 months.
  Group-1 consists of COPD patients whose have at least one fall (fallers)
  Interventions: Other: No intervention
- Group-2: The patients were classified based on the frequency of falls in the last 12 months.
  Group-2 consists of COPD patients whose have no history of falls (non-fallers).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention.

SUMMARY:
This cross-sectional study aims to investigate what daily activities increase the risk of falling in Chronic Obstructive Pulmonary Disease patients (COPD).

DETAILED DESCRIPTION:
To investigate the what daily activities increase the risk of falling in patients with COPD, twenty-eight voluntary patients with COPD, aged between 35-80 years will be divided into two groups: Group-1 have at least one fall (fallers) and Group-2 have no history of falls (non-fallers). Fall frequency will be investigated by asking patients to report any fall event in the last one month and the last 12-months. Assessments will be performed at baseline. Fear of falling will be assessed with Activities-Specific Balance Confidence (ABC) scale. Balance will be evaluated by Berg Balance Scale (BBS). The level of dyspnea during daily activities will be assessed with London Chest Activity of Daily Living (LCADL) scale. The global impacts of COPD symptoms on overall health status will be evaluated by The COPD Assessment Test (CAT). The Modified Medical Research Council Dyspnea (MMRC) scale and Six-Minute Walking Test (6MWT) will be used for evaluating the how dyspnea limits the patients' daily activities and functional capacity, respectively. Isometric muscle strength will be measured with a handheld dynamometer of quadriceps femoris. Pulmonary function data will be retrieved from the last 1-month clinical records of the COPD patients. Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 21.0. Among the groups, demographic and clinical variables will be compared with independent sample t-test for continuous variables and a chi-square test for categorical variables. The significance level will be set as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. stable disease (no severe exacerbations in the prior 3 months)
2. ability to walk independently
3. ability to read and write in Turkish
4. able to follow simple instructions
5. no pathology in visual ability and hearing

Exclusion Criteria:

1. a history of specific balance problems (i.e., diagnosed vestibular or neurological disorder)
2. severe musculoskeletal, neurological or cardiovascular disorders that limit mobility
3. use of medication(s) that may increase the risk of falls
4. participate in pulmonary rehabilitation in the lasts six months

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be patients with COPD diagnosed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines were recruited from Istanbul University, Department of Chest Diseases.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-08-31 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Activities-Specific Balance Confidence scale | Baseline
  Activities-Specific Balance Confidence (ABC) scale will be used for evaluating the confidence in maintaining the balance in activities daily living. It provides information on the level of concern about falls during16 community-based and home-based activities. Scale scores between 0 (unsafe) to 100 (completely safe) and the total score (0-1600) is divided by 16 to obtain an individual's ABC score, with higher scores indicating greater balance confidence. In patients with COPD, the ABC scale has demonstrated construct validity as well as criterion validity for falls. In addition, the participants will be also questioned concerning the occurrence of falls and the risk of falling during the activity in each item of the ABC scale.

SECONDARY OUTCOMES:
Fall frequency | Baseline
  Fall frequency will be investigated by asking patients to report any fall event in the last one month and the last 12-months. Participants will be asked: "Have you had any fall including a slip or trip in which you lost your balance and landed on the floor or ground or lower level?" Details about the circumstances of the fall and any resultant injury will be questioned.
Berg Balance Scale | Baseline
  Berg Balance Scale (BBS) will be used to assess the balance and determine the risk of falling in participants. It consists of 14-item evaluating a patient's ability to safely balance during a series of physical tasks. Scale scores between 0 (unable/unsafe) to 4 (independent/safe) and the total score ranges from 0 to 56, with higher scores indicating better balance control. The BBS has been demonstrated construct validity in patients with COPD.
London Chest Activity of Daily Living scale | Baseline
  London Chest Activity of Daily Living (LCADL) scale is used for assessing the level of dyspnea during daily activities. It is a 15-item scale comprised 4 domains: self-care (4 items), domestic (6 items), physical (2 items), and leisure (3 items). Each item scored between 0 (I wouldn't do it anyway) to 5 (I need help in doing this or someone to do it for me) and the total score ranges from 0 to 75, with higher scores indicating a more significant limitation in daily activities. The LCADL scale is a reliable, valid, and responsive instrument to assess limitations in performing daily activities in COPD patients. asked to rate each item in terms of risk of falling using a five-point scale, where 1=very low, 2=low, 3=moderate, 4=high, and 5=very high.
The COPD Assessment Test | Baseline
  The COPD Assessment Test (CAT) will be used for evaluating the global impacts of COPD symptoms on overall health status. Each item scores between 0 to 5 and the total score ranges from 0 to 40, with higher scores indicating the more severe impact of COPD on health status.
The strength of quadriceps femoris | Baseline
  The strength of quadriceps femoris of both sides will be measured with a hand-held dynamometer (kg.N-1) ''Nicholas Manual Muscle Tester" (model 01160, The Lafayette Instrument Company, Lafayette, Indiana). Each limb will assessed 3 times, with a recovery period of 30 seconds and the mean value will be calculated.
The Modified Medical Research Council Dyspnea scale | Baseline
  The Modified Medical Research Council Dyspnea (mMRC) scale will be used to determine how dyspnea limits the patients' daily activities performance. Itis a five-level rating scale consisting of just five items containing statements about the impact of dyspnea on the patients' daily activities performance and leading to a grade from 1 to 5. Higher scores indicate a greater impact of dyspnea on the patients' daily activities performance.
Six-Minute Walking Test (6MWT) | Baseline
  Six-Minute Walking Test (6MWT) is a reliable and valid test for evaluating functional capacity. Two 6MWTs will be performed according to the guidelines of the American Thoracic Society. The distance in meters covered over the 6 minutes of the test (6MWD) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)